CLINICAL TRIAL: NCT03863990
Title: Survival and Prognostic Factors in Pulmonary Arterial Hypertension. A Multicenter Observational Registry (START)
Brief Title: Study Performed at Various Medical Centers to Learn More About Survival and Expected Course of Pulmonary Arterial Hypertension, a Type of High Blood Pressure in the Lungs Related to the Narrowing of the Small Blood Vessels in the Lungs
Acronym: START
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20267
Record Dates: First submitted 2019-02-19; First posted 2019-03-05 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH prognosis; PAH outcomes; PAH survival; PAH risk status
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PAH: Adult male and female patients from Argentina diagnosed with pulmonary arterial hypertension (PAH) of WHO functional class I between 01-Jan-2012 and 31-Dec-2017 and with at least one year of follow-up.
  Interventions: Drug: PAH medication

INTERVENTIONS:
Drug: PAH medication — Any PAH-targeted medication

SUMMARY:
In this study researchers want to learn more about Pulmonary Arterial Hypertension, a type of high blood pressure in the lungs related to the narrowing of the small blood vessels in the lungs (group 1 according to WHO classification). Goal of the study is to describe the signs and risk factors of the illness at study start and the chances of survival.

DETAILED DESCRIPTION:
The primary objective of the study is to describe baseline clinical characteristics and overall survival in a cohort of patients with pulmonary arterial hypertension (PAH) of WHO functional class I in Argentina.

Secondary objectives are to study the discriminatory ability of the risk assessment tool presented in the European Society of Cardiology and European Respiratory Society (ESC/ERS) 2015 guidelines and to explore the potential prognostic advantage of a low-risk profile at follow-up as treatment goal.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive newly diagnosed patients by Right heart catheterization (RHC) from 01-Jan-2012 to 31-Dec-2017, belonging to one of the following of Group 1 PAH subgroups: Idiopathic (IPAH), or Heritable (HPAH), or Drug or toxin induced, or Associated (APAH) with one of the following: Connective tissue disease; Congenital heart disease with simple systemic to pulmonary shunt at least 1 year after surgical repair; Portal Hypertension or HIV infection.
* Diagnosis of PAH by RHC exhibiting a mean pulmonary artery pressure (MPAP) ≥ 25 mmHg and a pulmonary artery wedge pressure (PAWP) ≤15 mmHg at normal or reduced cardiac output, according to European Society of Cardiology and European Respiratory Society (ESC/ERS) 2009 guidelines or MPAP ≥ 25 mmHg and a PAWP ≤15 mmHg and a pulmonary vascular resistance (PVR) > 3 WU according to ESC/ERS 2015 guidelines.
* Patients with at least one year documented follow up or that have died or received transplant before 1 year of follow up after baseline RHC and that have initiated treatment with a PAH-targeted medication.

Exclusion Criteria:

* Patients with severe concomitant left heart disease (left ventricular ejection fraction <35%).
* Patients with restrictive lung disease (Forced vital capacity (FVC) <60% predicted) other than connective tissue disease or obstructive lung disease (forced expiratory volume (FEV) <60% predicted, with FEV1/FVC<70%).
* Clinical or radiological evidence of Pulmo-Veno-Occlusive Disease (PVOD) or Pulmonary Capillary Haemangiomatosis (PCH).
* Hypertrophic obstructive cardiomyopathy.
* Severe proven or suspected coronary artery disease.
* Congenital or acquired valvular or myocardial disease if clinically significant apart from tricuspid valvular insufficiency due to pulmonary hypertension.
* Underlying medical disorders at baseline with an anticipated life expectancy below 2 years (e.g. active cancer disease with localized and/or metastasized tumor mass) or Clinical relevant hepatic dysfunction (Child-Pugh B and C) or Renal insufficiency (glomerular filtration rate <30 mL/min).
* Diagnosis of a pulmonary hypertension from WHO groups 2, 3, 4 or 5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with pulmonary arterial hypertension from tertiary care centers in Argentina
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Age at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Sex | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Ethnicity | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Descriptive analysis of comorbidities at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
PAH-subgroup at baseline as assessed by physician | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  PAH-subgroups may be idiopathic, heritable, drug- or toxin-induced, or associated PAH (with CTD or HIV or portopulmonary hypertension or repaired congenital heart disease).
Right atrial pressure at baseline by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary artery pressure at baseline by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary vascular resistance at baseline by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary artery wedge pressure (PAWP) at baseline by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Cardiac Index (CI) at baseline by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Mixed venous oxygen saturation (SvO2) at baseline by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary vasoreactivity at baseline by pulmonary artery pressure | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Yes / No - variable
Peak oxygen consumption by cardiopulmonary exercise test at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Right atrial area at baseline by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pericardial effusion at baseline by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Patients may have no, mild, moderate or severe pericardial effusion.
Right ventricular function at baseline by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Patients may have a normal, mild, moderate and severe right ventricular function.
Tricuspid annular plane systolic excursion (TAPSE) at baseline by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary artery systolic pressure at baseline by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Left ventricular ejection fraction at baseline by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
6-minute walking distance at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary hypertension functional class according to WHO classification at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Four functional classes ranging from Class I (Pulmonary hypertension without limited physical activity) to Class IV (Pulmonary hypertension with strongly limited physical activity).
Time from onset of diagnostic symptoms to PAH-diagnosis | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Symptoms progression at baseline assessed by physician | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Patient may display no, a slow or rapid progression of symptoms.
Syncope frequency at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  No, occasional or repeated syncope
Systolic blood pressure at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Heart rate at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Body weight at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Body height at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Body mass index at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Concentration of diagnostic markers for heart failure in blood at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Used diagnostic marker are either Brain natriuretic Peptide (BNP) or N-terminal pro b-type Natriuretic Peptide (NT-proBNP).
Drug class of supportive PAH treatment | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Supportive treatments for PAH are assigned to four drug classes: diuretics, anticoagulants, oxygen and other.
Drug class of PAH-treatment after diagnosis | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  PAH-treatments are assigned to six drug classes: endothelin receptor antagonists (ERA), PDE5 inhibitors, prostanoides, prostacyclin receptor agonists, soluble guanylate cyclase (sGC) stimulants and calcium blockers.
PAH risk status at baseline according to ESC/ERS 2015 guidelines | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Patients may have a low, intermediate or high risk for PAH according to the European Society of Cardiology and European Respiratory Society 2015 guidelines.
Overall survival rate | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Time from diagnosis to death from any cause | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018

SECONDARY OUTCOMES:
Right atrial pressure at follow-up by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary artery pressure at follow-up by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary vascular resistance at follow-up by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary artery wedge pressure (PAWP) at follow-up by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Cardiac Index (CI) at follow-up by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Mixed venous oxygen saturation (SvO2) at follow-up by right heart catheterization hemodynamics | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Peak oxygen consumption by cardiopulmonary exercise test at follow-up | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Right atrial area at follow-up by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pericardial effusion at follow-up by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Right ventricular function at follow-up by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Tricuspid annular plane systolic excursion (TAPSE) at follow-up by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary artery systolic pressure at follow-up by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Left ventricular ejection fraction at follow-up by echocardiography | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
6-minute walking distance at follow-up | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary hypertension functional class according to WHO classification at baseline | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Four functional classes ranging from Class I (Pulmonary hypertension without limited physical activity) to Class IV (Pulmonary hypertension with strongly limited physical activity).
Symptoms progression at follow-up | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Syncope frequency at follow-up | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Concentration of diagnostic markers for heart failure in blood at follow-up | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Used diagnostic marker are either Brain natriuretic Peptide (BNP) or N-terminal pro b-type Natriuretic Peptide (NT-proBNP).
PAH risk status at follow-up according to ESC/ERS 2015 guidelines | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Patients may have low, intermediate and high risk for PAH according to the European Society of Cardiology and European Respiratory Society 2015 guidelines.
Cause of death | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Time from diagnosis to death from any cause | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Pulmonary transplant | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Yes or No
Time from diagnosis to pulmonary transplant | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Time from diagnosis to first hospitalization due to PAH-progression | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Number of hospitalizations per year due to PAH-progression | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Proportion of patients with low PAH risk | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Risk status is assessed according to the Society of Cardiology and European Respiratory Society (ESC/ERS) 2015 guidelines.
Proportion of patients with intermediate+high PAH risk | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Risk status is assessed according to the Society of Cardiology and European Respiratory Society (ESC/ERS) 2015 guidelines.
Survival rate of patients with low risk for PAH | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
Survival rate of patients with intermediate or high risk for PAH | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
PAH risk status of patients without transplant being alive at the date of latest medical records according to ESC/ERS 2015 guidelines | Retrospective analysis of data from 01-Jan-2012 to 31-Dec-2018
  Patients may have low, intermediate and high risk for PAH according to the European Society of Cardiology and European Respiratory Society 2015 guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Many facilities, Multiple Locations, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/